CLINICAL TRIAL: NCT03109522
Title: A Pilot Randomized Controlled Trial Comparing the Axillary Reverse Mapping (ARM) Technique to Standard Axillary Surgery in Breast Cancer Patients.
Brief Title: Axillary Reverse Mapping (ARM) Technique
Acronym: ARM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Peter Lovrics, Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TR-182
Record Dates: First submitted 2016-10-27; First posted 2017-04-12 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Invasive Breast Cancer; Ductal Carcinoma in Situ of the Breast
Keywords: axillary reverse mapping (ARM); sentinel lymph node biopsy (SLNB); axillary lymph node dissection (ALND); lymphedema; breast cancer; surgery
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Lymphedema; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- axillary reverse mapping (Experimental): Axillary reverse mapping and sentinel lymph node biopsy (ARM/SLNB) or Axillary reverse mapping and axillary lymph node dissection (ARM/ALND)
  Interventions: Procedure: axillary reverse mapping (ARM)
- standard axillary surgery (Active Comparator): The control group will have standard sentinel lymph node biopsy (SLNB) or axillary lymph node dissection (ALND) without identifying or sparing upper-limb lymphatics and nodes (blue dye is not injected).
  Interventions: Procedure: Standard axillary surgery (SLNB or ALND)

INTERVENTIONS:
Procedure: axillary reverse mapping (ARM) — ARM/SLNB: patient will be injected with technetium-99 radiolabelled colloid (Tc-99) into the subareolar area of breast, then 1-2 mls of blue dye (patent blue dye) injected subcutaneously into the medial ipsilateral arm, just proximal to the medial epicondyle of the elbow, at the start of the surgical procedure. the SLN(s) will be identified ("hot node") and removed, and any blue lymph nodes and lymphatics will be preserved intact, and only removed or disrupted if there is 'crossover" (i.e. the blue node is also the SLN) or if clinically suspicious for metastatic disease. ARM/ALND: 1-2 mls of blue dye will be injected subcutaneously into the medial ipsilateral arm at the start of the surgical procedure. Surgeons will perform a standard level I and II axillary dissection and any blue lymph nodes or lymphatics will be preserved intact, and only removed or disrupted if blue nodes are suspicious for metastatic disease.
  Arms: axillary reverse mapping
Procedure: Standard axillary surgery (SLNB or ALND) — The control group will have standard SLNB or ALND surgery without identifying or sparing upper-limb lymphatics and nodes (blue dye is not injected).
  Arms: standard axillary surgery

SUMMARY:
The purpose of this pilot study is to compare a new surgical technique (axillary reverse mapping) to standard axillary surgery in patients diagnosed with invasive or in situ breast cancer.

DETAILED DESCRIPTION:
Lymphedema is a major chronic morbidity that occurs in patients undergoing treatment for breast cancer (BC). Surgery for BC includes axillary surgery with either sentinel lymph node biopsy (SLNB) or axillary lymph node dissection (ALND). Lymphedema occurs due to removal or disruption of lymphatic drainage of the arm that overlaps with drainage of the breast. The risk of lymphedema increases significantly with adjuvant radiation. Axillary reverse mapping (ARM) is a technique where blue dye is injected into the upper arm at surgery, allowing direct visualization of arm lymphatics and nodes during either SLNB or ALND. This allows preservation of arm lymphatics unless there is suspicion of metastatic disease in ARM lymphatics or if the ARM node is/are also the sentinel lymph node. Studies to date have largely been observational cohort studies, and mainly with low risk patients undergoing SLNB only. There is only one published randomized controlled trial, and this included only patients undergoing modified radical mastectomy.Our proposal is a prospective randomized pilot study. The study population includes patients undergoing axillary surgery (SLNB with mastectomy or ALND with either BCS or mastectomy or completion ALND after positive SLNB). The intervention group will undergo ARM; the control will undergo standard surgical treatment. Both groups will undergo standardized baseline and postoperative arm measurements and patients will complete symptom and quality of life questionnaires. The purpose is to determine the feasibility of the ARM technique, its accuracy in identifying and sparing arm lymphatics, and its ability to reduce the risk of lymphedema.

ELIGIBILITY:
Inclusion Criteria: women diagnosed with invasive breast cancer or ductal carcinoma in situ receiving the following treatment:

1. mastectomy and sentinel lymph node biopsy
2. breast conserving surgery or mastectomy and axillary lymph node dissection
3. completion axillary lymph node dissection after positive sentinel lymph node biopsy
4. cases receiving neo-adjuvant therapy (chemotherapy or hormonal therapy) who are having axillary lymph node dissection as part of their surgical treatment -

Exclusion Criteria:

1. males with breast cancer
2. women less than 18 years of age
3. known allergic reaction to patent blue dye
4. pregnant
5. previous radiation therapy to affected side
6. clinical N2/N3 disease -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Lymphedema | Change from baseline to 6 months post-operative
  Arm circumference measurements of both arms. An arm volume difference of > 10% will be considered clinically significant lymphedema
Lymphedema | Change from baseline to 12 months post-operative
  Arm circumference measurements of both arms. An arm volume difference of > 10% will be considered clinically significant lymphedema

SECONDARY OUTCOMES:
EORTC-QLQ-C30 | Change from baseline to 6 months post-operative
  General quality of life
EORTC-QLQ-C30 | Change from baseline to 12 months post-operative
  General quality of life
Disabilities of the Arm and Shoulder and Hand (DASH) | Change from baseline to 6 months post-operative
  arm symptoms and disabilities
Disabilities of the Arm and Shoulder and Hand (DASH) | Change from baseline to 12 months post-operative
  arm symptoms and disabilities
Post-operative complications | 30 days post-op
  infection, hematoma, problems with wound healing
Breast Cancer and Lymphedema Symptom Experience Index (BCLE-SEI) Part 1 | Change from baseline to 6 months post-operative
  arm symptoms and pain
Breast Cancer and Lymphedema Symptom Experience Index (BCLE-SEI) Part 1 | Change from baseline to 12 months post-operative
  arm symptoms and pain

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lovrics, MD, Principal Investigator — McMaster University; Nicole Hodgson, MD, MSc, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Juravinski Hospital and Cancer Centre, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No